CLINICAL TRIAL: NCT07016035
Title: Translation and Validation of the French Version of the Health-related Quality of Life Questionnaire for the Polycystic Ovary Syndrome: the mPCOSQ-F.
Brief Title: Translation and Validation of the French mPCOSQ (mPCOSQ-F).
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PS25052
Record Dates: First submitted 2025-05-13; First posted 2025-06-11 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome Health-related Quality of Life
Keywords: polycystic ovary syndrome; PCOS; quality of life; health-related quality of life; mPCOSQ; questionnaire; SF-36; French
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Polycystic ovary syndrome: patients with Polycystic ovary syndrome
  Interventions: Other: mPCOSQ-F and SF-36

INTERVENTIONS:
Other: mPCOSQ-F and SF-36 — Questionnaires

SUMMARY:
This study is a prospective, observational, bicentric study, evaluating the validity and reliability of a French version of the mPCOSQ questionnaire (mPCOSQ-F), used to assess health-related quality of life (HRQOL) in women with polycystic ovary syndrome.

The first stage of the study consisted in translating the questionnaire from English to French.

Patients agreeing to take part in the study will complete the mPCOSQ-F and the SF-36 (generic HRQOL questionnaire). After 1 to 2 weeks, patients will receive the mPCOSQ-F and complete it again.

DETAILED DESCRIPTION:
The aim of this study is to assess the validity and reliability of a French version of the mPCOSQ questionnaire (mPCOSQ-F), used to assess health-related quality of life (HRQOL) in women with polycystic ovary syndrome.

Women aged 18 to 45 years with a diagnosis of polycystic ovary syndrome will be included.

The first stage of the study consisted in translating the questionnaire from English to French.

Patients agreeing to take part in the study will complete the mPCOSQ-F and the SF-36 (generic HRQOL questionnaire). After 1 to 2 weeks, patients will receive the mPCOSQ-F and complete it again.

The pre-test phase purpose is to appraise the face validity and feasibility of the questionnaire through phone interviews with the thirty first respondents.

In the final phase, we aimed to evaluate the validity and reliability of the mPCOSQ, and to compare it to the SF-36.

ELIGIBILITY:
Inclusion criteria:

* Women aged 18 to 45
* Fluent in french
* Having a diagnosis of PCOS according to the international recommendations published in 2023
* Willing to participate in the study
* Affiliated to the french social security system

Exclusion criteria:

* Diagnosis of adrenal hyperplasia, androgen-producing tumor, Cushing's syndrome, or thyroid disorder
* Pregnancy or breast-feeding
* Under legal protection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients were PCOS women recruited from the Reims University Hospital and the Charleville-Mézières Hospital when presenting to endocrinology, gynaecology or reproductive medicine consults.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Content validity of mPCOSQ as determined by the experts group | At 2 years
Feasibility of mPCOSQ | At 2 years
Acceptability of mPCOSQ | At 2 years
Structure validity of mPCOSQ | At 2 years
Reproductibility of mPCOSQ | At 2 years
Reliabilty of mPCOSQ | At 2 years
Total mPCSOQ score | At 15 days
SF-36 scores | At 1 day
Scores in the " weight " domain based on BMI | At 1 day
Scores in the " fertility " domain based on the need for reproductive medicine or parenthood | At 1 day
Scores in the " hirsutism " domain based on the Ferriman-Gallwey score | At 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France